CLINICAL TRIAL: NCT04253678
Title: Vortioxetine for Cancer Patients With Depression: An Observational Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Dr Ng Chong Guan, Associate Professor, University of Malaya
Other Study IDs: VOR001
Record Dates: First submitted 2020-01-28; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Major Depressive Disorder; Cancer
Keywords: depression; cancer; vortioxetine; cognition; quality of life; antidepressant
MeSH Terms: conditions — Depressive Disorder, Major; Neoplasms; Depression | interventions — Vortioxetine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study group: Study participants will be started on a flexible-dose of vortioxetine (5-20 mg) followed by a baseline assessment of primary outcomes using the Montgomery-Asberg Depression Rating Scale (MADRS) and the Perceived Deficit Questionnaire - 5 items (PDQ-5), and secondary outcomes using the EORTC Quality of life Questionnaire (QLQ-C30) and Clinical Global Impression (CGI). The assessment timelines will be at week 2, week 4, week 8, and week 12.
  Side effects, if any, will be recorded using the Antidepressant Side-effect Checklist (ASEC).
  Interventions: Drug: Vortioxetine

INTERVENTIONS:
Drug: Vortioxetine — Flexible dosing from 5mg to 20mg based on attending psychiatrist's discretion
  Other Names: Brintellix

SUMMARY:
The purpose of this observational antidepressant study is to determine the efficacy of vortioxetine on depression and cognitive function, and elucidate its potential effects on quality of life in patients with cancer (of any origin). We hypothesise that given its unique mechanism of action as a multimodal serotonin modulator, vortioxetine is set to achieve the above goals while maintaining a favourable side effect profile.

DETAILED DESCRIPTION:
Cancer is always a feared illness and the diagnosis of cancer has huge psychological impact on the patients. Depression is one of the most common psychiatric sequelae and affects the disease outcome in cancer patients. Along with depression, cancer patients are also vulnerable to develop cognitive impairment. It could be related to the cancer or its treatment. Cognitive impairment that occurs among cancer patient is known as cancer related cognitive impairment (CRCI). Depression together with cognitive impairment adversely affect the quality of life of cancer patients. To date, the optimal treatment of depression in cancer is not established. The number of studies investigated the efficacy of pharmacotherapy for depression in cancer patient is limited. The evidence of treatment for cognitive impairment in depressed cancer patients is even more scarce.

Vortioxetine is one of the latest marketed antidepressants in Malaysia. It has numerous additional effects as compared to other conventional antidepressants. In addition to blockade of the serotonin transporter (SERT), vortioxetine has affinity for 5-HT1A, 5-HT1B, 5-HT3, and 5-HT7 receptors and as such, it is described as a 'multimodal serotonin modulator'. This may explain the additional benefit of vortioxetine in the treatment of depression as compared to other antidepressants. Furthermore, the unique mechanism of action of vortioxetine was also reported to improve cognitive function in patients with depression.

General Objective:

To examine the effect of vortioxetine in improving the depressive symptoms, cognitive impairment and quality of life in cancer patients who have major depressive disorder.

Specific Objectives:

1. To determine whether treatment with antidepressant vortioxetine is effective to improve depressive symptoms in patients diagnosed with cancer (of any origin) and major depressive disorder.
2. To determine whether treatment with antidepressant vortioxetine is effective to improve cognitive impairment in patients diagnosed with cancer (of any origin) and major depressive disorder.
3. To determine whether treatment with antidepressant vortioxetine is effective to improve quality of life in patients diagnosed with cancer (of any origin) and major depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years old
* Literate and able to understand English or Malay
* Diagnosed with Major Depressive Disorder
* Diagnosed with cancer of any origin

Exclusion Criteria:

* Medically unstable
* Delirium
* Actively psychotic
* Cognitive deficits of other causes
* Primary or secondary cerebral/cranial tumors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cancer of any origin who are diagnosed with Major Depressive Disorder based on DSM 5 will be screened for the study. Those consented will be enrolled in the observational study. The total target sample size will be 140 subjects. The study will be conducted at the psychiatric clinic (Psycho-oncology clinic on every Thursday) in University Malaya Medical Centre as a main centre as well as other centres in Malaysia.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2019-12-12 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Changes in Montgomery-Asberg Depression Rating Scale (MADRS) | baseline (week 1), week 2, week 4, week 8, week 12
  The MADRS is a widely used clinical rating scale for depression. It consists of 10 items evaluating core symptoms of depression (Montgomery & Äsberg, 1979; Montgomery et al., 1978). Nine of the items are based upon patient report, and one is on the rater's observation during the rating interview. MADRS items are rated on a 0-6 continuum (0=no abnormality, 6=severe). The MADRS is relatively quick to administer and addresses core mood symptoms of depression such as sadness, tension, lassitude, pessimistic thoughts, and suicidal thoughts.
Changes in Perceived Deficits Questionnaire - 5 items (PDQ-5) | baseline (week 1), week 2, week 4, week 8, week 12
  The PDQ-5 is a brief patient-rated scale to assess subjective cognitive dysfunction in people with depression. The PDQ originally is a 20-item questionnaire developed by Dr. Michael Sullivan at McGill University as a scale for use in patients with multiple sclerosis that generates a total score and 4 subscale scores (attention/concentration, retrospective memory, prospective memory, and planning/organization) (Sullivan et al., 1990). A 5-item version (PDQ-D-5) is a brief version and has been adapted and validated for use in patients with major depressive disorder.

SECONDARY OUTCOMES:
Changes in Clinical Global Impression (CGI) | baseline (week 1), week 2, week 4, week 8, week 12
  The CGI allows psychiatrist to assess the patient's condition relative to baseline and rate the change on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse).
Changes in EORTC-QLQ-C30 | baseline (week 1), week 2, week 4, week 8, week 12
  The EORTC QLQ-C30 is widely used clinical scale for measurement of cancer-specific quality of life. It contains five functioning scales (physical, social, role, cognitive, and emotional functioning), eight symptom scales (fatigue, nausea/vomiting, pain, dyspnea, sleep disturbances, appetite loss, constipation, and diarrhea), financial impact, and overall quality of life. All scale scores are linearly converted to range from 0 to 100. For the functioning scales and global QOL higher scores indicate better functioning; for the symptom scales higher scores indicate higher symptom burden (Aaronson et al., 1993).

CONTACTS AND LOCATIONS:
Overall Officials: Chong Guan Ng, Principal Investigator — UMMC
Locations (8):
- Malaysia (8):
  - Hospital Raja Permaisuri Bainun, Ipoh, Ipoh, Perak
  - Hospital Tengku Ampuan Rahimah Klang, Klang, Selangor
  - Hospital Sungai Buloh, Sungai Buloh, Selangor
  - National Cancer Institute, Kuala Lumpur
  - Hospital Kuala Lumpur, Kuala Lumpur
  - Pusat Perubatan Universiti Kebangsaan Malaysia, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Putrajaya, Kuala Lumpur

IPD SHARING:
Plan to Share IPD: No